CLINICAL TRIAL: NCT04440618
Title: Prevalence of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) Following Squamous Cell Carcinomas of the Oropharynx Treatment by Combined Chemoradiotherapy
Acronym: COROSAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COROSAS
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea-hypopnea; Oropharyngeal Cancer
Keywords: combined chemoradiotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study's aim is to determinate the prevalence of obstructive sleep apnea hypopnea syndrome after treatment by combined chemoradiotherapy in a locally advanced stages treated population of oropharyngeal cancer. Indeed, the level of knowledge about the consequences of oropharyngeal cancer treatment on sleep quality remains poor but the few studies published on the subject suggest an increased risk of development of OSAHS for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Performance Status 0-2
* Squamous cell carcinoma of the oropharynx treated with concomitant chemoradiotherapy
* Treatment termination time greater than 6 months at inclusion
* Tumor classification (American Joint Committee on Cancer 8th) T2-T4 N0-N3
* Patient in complete remission at inclusion
* patient's consent's obtained after information

Exclusion Criteria:

* Previous treatment for upper aerodigestive tract cancer
* Incomplete radiotherapyTreatment
* Neurological pathology wich may affect the functions of the upper aerodigestive tract
* Pregnant or breastfeeding woman
* Unweaned alcoholism
* Tracheotomized patient at the time of the study
* Patient under protection: subjects with guardianship or under law protection
* No health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disease-free patients treated for locally advanced oropharyngeal cancer for over 6 months by radio-chemotherapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea hypopnea syndrome after treatment by combined chemoradiotherapy. | Day 28
  Number of patients with obstructive sleep apnea hypopnea syndrome after treatment combined chemoradiotherapy.

SECONDARY OUTCOMES:
Severity of OSAHS as a function of the post-therapeutic delay. | Day 28
  Value of the AHI as a function of the post-therapeutic delay which corresponds to the delay compared to the end of the curative treatment carried out for squamous cell carcinoma of the oropharynx. It is obtained after the inclusion visit and the realization of the polygraphy with the IAH score. OSAHS is mild (if IAH ≥ 5 / h and <15 / h), moderate (if IAH ≥ 15 / h and ≤ 30 / h) or severe (if IAH> 30 / h)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France